CLINICAL TRIAL: NCT00580866
Title: Multi-Center Controlled Trial of Static Progressive Splinting Status Post Elbow Fractures and Dislocations
Brief Title: Progressive Splinting Status Post Elbow Fractures and Dislocations
Acronym: JAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, William Obremskey, Associate Professor, Vanderbilt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 051196
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Upper Extremity Fracture; Upper Extremity Dislocation; Fractures, Comminuted; Elbow Fracture; Elbow Dislocation
Keywords: Elbow; Upper Extremity Fractures; Distal Humerus; Elbow Injuries; Dislocations; Peri-articular Elbow Injuries
MeSH Terms: conditions — Fractures, Comminuted; Elbow Fractures; Elbow Injuries; Joint Dislocations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Joint Active Systems Brace (JAS Brace) (Experimental): Elbow is placed in a brace to apply an extension force
  Interventions: Device: JAS Brace
- PT Only Group (No Intervention): No brace is used

INTERVENTIONS:
Device: JAS Brace — For approximately 6 weeks after surgery, the brace will be utilized for a period of 30 minutes, 3 times per day. Participants will also receive physical therapy 3 times per week.
  Other Names: JAS Static Progressive Stretch; Joint Active Systems Brace (JAS Brace); Static Stretching Brace; Static Progressive Stretching Brace
  Arms: Joint Active Systems Brace (JAS Brace)

SUMMARY:
The purpose of this study is to help determine if a static stretching brace in addition to physical therapy decreases the incidence of secondary operations, increases range of motion, and individual patient function.

DETAILED DESCRIPTION:
Fractures and dislocations about the elbow are high energy injuries which are often comminuted and associated with extensive soft tissue damage and are very difficult to treat. The most problematic complication for these fractures is the potential development of a cosmetic defect and functional disability due to the loss of 20 degrees to 30 degrees of terminal extension of the elbow. It has been found imperative that early motion and physical therapy be implemented to help produce the best results in terms of a patient's range of motion and decreases secondary surgeries.

We intend to examine a group of patients with distal humerus and elbow fracture/dislocations who use static stretching braces along with physical therapy (PT) within 3 weeks after surgery, in contrast to physical therapy treatment alone after surgery. The static stretching brace group will have a small electronic circuit attached to the brace that will record patient's usage.

Improvement of patient's overall functional outcome will also be measured by a standard functional outcome instrument, the Disabilities of Arm, Shoulder and Hand (DASH) form. The DASH Form is a standard functional outcome instrument specific to upper extremity injuries. In addition, a more general measure, the Visual Analog Scale (VAS), will be used to assess pain.

The use of the static motion brace may help eliminate the necessity of additional treatments, saving both pain and suffering, as well as monetary costs for the patient, while simultaneously producing a better long term functional and cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Extra or intraarticular distal humerus or elbow fracture or fracture/dislocation
* Agrees to participate and signs informed consent
* English Speaking (outcome questionnaires are validated for English only)

Exclusion Criteria:

* Less than 18 years of age
* Closed Head Injury
* Burn Injuries
* Ipsilateral upper extremity fracture(s) requiring surgery
* Nonunion of prior distal humerus fracture or fracture dislocation
* Type 3 open distal humerus fracture dislocation
* Insufficient fracture fixation to allow early range of motion
* Transient population with no fixed address
* Not willing to sign informed consent
* Does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Obremskey, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Orthopaedic Institute, Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Brace Group: JAS Brace: For approximately 6 weeks after surgery, the brace will be utilized for a period of 30 minutes, 3 times per day. Participants will also receive physical therapy 3 times per week.
Period: Overall Study
Arm/Group | Brace Group | PT Only Group
Started | 10 | 7
Completed | 8 | 5
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brace Group | PT Only Group | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Elbow ROM at 12 Months
Description: The goal of this study is to determine if static progressive splinting eliminates deformity by improving patients' range of motion.
Time Frame: 2 weeks, 6 weeks, 3 months, 6 months, 12 months post-operatively
Population: Elbow ROM at 12 months analysis. Data was not collected at 2 weeks, 6 weeks, 3 months, 6 months due to poor enrollment.
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Brace Group | PT Only Group
Number analyzed (Participants) | 8 | 5
degrees | 121 [110 to 130] | 123 [119 to 129]

2. Secondary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH) Score
Description: Improvement of patient's overall functional outcome will be measured by a standard functional outcome instrument, the DASH Score. The results can range from 0 (no disability) to 100 (worst )
Time Frame: 12 months post-operatively
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Brace Group | PT Only Group
Number analyzed (Participants) | 8 | 5
scores on a scale | 25 [21 to 29] | 23 [19 to 27]

ADVERSE EVENTS:
Arm/Group | Brace Group | PT Only Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No